CLINICAL TRIAL: NCT02277561
Title: Prediction of Response of Brain Metastases to Brain Irradiation Using Voxel Based Diffusion Tensor Imaging
Brief Title: Voxel Based Diffusion Tensor Imaging in Predicting Response in Patients With Brain Metastases Undergoing Whole Brain Radiation Therapy or Stereotactic Radiosurgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB approved but never implemented
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Madhur Garg, Principal Investigator, Albert Einstein College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-01-047; NCI-2014-01015 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13-01-047 (Other: Albert Einstein College of Medicine); P30CA013330 (NIH)
Record Dates: First submitted 2014-10-27; First posted 2014-10-29 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Tumors Metastatic to Brain; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Brain Neoplasms | interventions — Diffusion Tensor Imaging; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

ARMS (1):
- Diagnostic (VB-DTI, MRI) (Experimental): Patients undergoing WBRT for a total of 10 fractions also undergo VB-DTI MRI at baseline, 1 week after WBRT initiation, and 7-11 days after completion of WBRT. Patients undergoing SRS without WBRT also undergo VB-DTI MRI at baseline and 7-11 days after completion of SRS.
  Interventions: Procedure: diffusion tensor imaging; Radiation: whole-brain radiation therapy; Radiation: stereotactic radiosurgery; Procedure: contrast-enhanced magnetic resonance imaging; Procedure: diffusion-weighted magnetic resonance imaging

INTERVENTIONS:
Procedure: diffusion tensor imaging — Undergo VB-DTI
Radiation: whole-brain radiation therapy — Undergo WBRT
  Other Names: WBRT; whole-brain radiotherapy
Radiation: stereotactic radiosurgery — Undergo SRS
Procedure: contrast-enhanced magnetic resonance imaging — Undergo contrast-enhanced MRI
  Other Names: Contrast-enhanced MRI
Procedure: diffusion-weighted magnetic resonance imaging — Undergo DW MRI
  Other Names: diffusion-weighted MRI

SUMMARY:
This pilot clinical trial studies how well voxel based diffusion tensor imaging in predicting response in patients with brain metastases undergoing whole-brain radiation therapy or stereotactic radiosurgery. Voxel based diffusion tensor imaging (VB-DTI) may allow doctors to measure response to whole brain radiation therapy or stereotactic radiosurgery earlier than is possible with a standard magnetic resonance imaging. The earlier ability to measure response may allow for consideration of alternative therapies at an earlier stage.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if voxel based diffusion tensor imaging will provide an early predictive assessment of therapy response, as compared to radiographic volumetric response criteria.

OUTLINE:

Patients undergoing whole-brain radiation therapy (WBRT) for a total of 10 fractions also undergo VB-DTI magnetic resonance imaging (MRI) at baseline, 1 week after WBRT initiation, and 7-11 days after completion of WBRT. Patients undergoing stereotactic radiosurgery (SRS) without WBRT also undergo VB-DTI MRI at baseline and 7-11 days after completion of SRS.

After completion of study, patients are followed up every 2 months for 6 months and then every 6 months until death.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple lesions from solid tumors on clinical MRI diagnosing the brain metastases may be treated with either WBRT or SRS if clinically indicated at the time of presentation but not both
* Karnofsky performance status (KPS) >= 70
* Patients presenting with brain metastases from a newly diagnosed cancer may have systemic disease (brain disease at the time of initial cancer diagnosis)
* Patients with a history of cancer, but newly diagnosed brain metastases must have clinically stable systemic disease
* If a biopsy is performed, the patient has to be at least 1 week post-biopsy
* The patient must be able to commit to diffusion-weighted magnetic resonance (MR) imaging, diffusion tensor imaging (DTI), and chemical shift imaging (CSI) prior to treatment, after the first week of treatment, and 7-11 days after the completion of treatment at the Magnetic Resonance Research Center (MRRC)
* Patients undergoing SRS without WBRT must be able to commit to diffusion-weighted MR imaging, DTI, and CSI prior to treatment, and 7-11 days after the completion of the SRS treatment at the MRRC
* The patient must also be able to commit to post-treatment follow-up visits at Montefiore Medical Center involving serial MR imaging; the follow-up visits are to occur bimonthly for 6 months and then every 6 months until death

Exclusion Criteria:

* Any medical condition, which would make the imaging studies or WBRT unsafe or poorly tolerated
* Patient is receiving concurrent chemotherapy
* Known allergic reaction to contrast or shellfish
* Patients with brain metastases to be treated with radiosurgery
* Patients with brain metastasis resulting from hematologic malignancies and small cell lung cancer
* Implanted metal devices or foreign bodies that serve as a contraindication to MR imaging
* Creatinine > 1.4 mg/dl and creatinine clearance < 20 mg/dl
* Uncontrolled, clinically significant cardiac arrhythmias
* Severe claustrophobia
* Pregnant female
* Any prior radiation therapy to the brain
* KPS < 70
* Patients with leptomeningeal disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Percentage of voxel-based mean apparent diffusion coefficient (ADC) increase per lesion | Up to 3 years
Volume fraction of voxels showing treatment-related VB-DTI changes for each lesion | At 4 months
  Spearman's rank analysis will be used to determine if a correlation exists between the volume fraction of voxels showing treatment-related VB-DTI changes and the volumetric radiographic response for each lesion. Statistical significance will be achieved with a p value < 0.05.
Volumetric radiographic response for each lesion | At 4 months
  Spearman's rank analysis will be used to determine if a correlation exists between the volume fraction of voxels showing treatment-related VB-DTI changes and the volumetric radiographic response for each lesion. Statistical significance will be achieved with a p value < 0.05. Statistical significance will be achieved with a p value < 0.05.
Change in a lesion's overall mean ADC | Baseline to 4 months
  Spearman's rank analysis will be used to determine if a correlation exists between the volume fraction of voxels showing treatment-related VB-DTI changes and the volumetric radiographic response for each lesion. Statistical significance will be achieved with a p value < 0.05. Statistical significance will be achieved with a p value < 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Madhur Garg, Principal Investigator — Montefiore Medical Center
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States